CLINICAL TRIAL: NCT06605950
Title: A 2-Part, Phase 1, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Doses of Dual-burst Release of Xanomeline With Immediate-Release Trospium Chloride Versus KarXT in Healthy Adult and Elderly Participants of Japanese Ethnicity (Part 1) and an Open-label Study to Assess the Effect of Omeprazole on the Pharmacokinetics of Dual-burst Release of Xanomeline With Immediate-Release Trospium Chloride in Healthy Adult Participants (Part 2)
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics (PK) of Xanomeline With Trospium Chloride Versus KarXT in Healthy Adult and Elderly Participants of Japanese Ethnicity and to Assess the Effect of Omeprazole on the PK of Xanomeline With Trospium Chloride in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0030
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: Japanese; Elderly; Adult; Healthy; Pharmacokinetics; BMS-986510; BMS-986519; KarXT; Omeprazole; Drug interaction
MeSH Terms: interventions — xanomeline; trospium chloride; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 of this study is double-blind while Part 2 is open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental)
  Interventions: Drug: KarXT; Drug: Placebo
- Group B (Experimental)
  Interventions: Drug: KarXT; Drug: Placebo
- Group C (Experimental)
  Interventions: Drug: KarXT; Drug: KarX-EC; Drug: Placebo
- Group D (Experimental)
  Interventions: Drug: KarXT; Drug: KarX-EC; Drug: Omeprazole

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510; Xanomeline/Trospium Chloride
Drug: KarX-EC — Specified dose on specified days
  Other Names: BMS-986519; Xanomeline Enteric-coated
  Arms: Group C; Group D
Drug: Placebo — Specified dose on specified days
  Arms: Group A; Group B; Group C
Drug: Omeprazole — Specified dose on specified days
  Arms: Group D

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics (PK) of multiple doses of KarXT + KarX-EC capsules versus KarXT capsules in healthy adult and elderly participants of Japanese ethnicity and to assess the effect of multiple doses of omeprazole on the exposure of xanomeline and trospium administered as KarXT + KarX-EC capsules in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria

* Inclusion Criteria for Healthy Adult Japanese Participants (Group A):.
* Healthy adult participants must be 19 to 55 years of age, inclusive.

  i) Both participant's biological parents are of ethnic Japanese ancestry. Participants must be first generation Japanese.

ii) Must have a body mass index (BMI) of 18.0 to 32.0 kg/m2 (inclusive), at the time of signing the ICF.

iii) Must have an estimated glomerular filtration rate (eGFR) of ≥ 90 mL/min/1.73m2 by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at the screening visit. One repeat measurement is allowed.

* Inclusion Criteria for Healthy Elderly Japanese Participants (Groups B and C):.
* Healthy elderly participants must be 56 to 90 years of age, inclusive.

  i) Both participant's biological parents are of ethnic Japanese ancestry. Participants must be first generation Japanese.

ii) Must have a BMI ≥ 18.0 and ≤ 35.0 kg/m2 (inclusive), at the time of signing the ICF.

iii) Must have an eGFR of > 60 mL/min/1.73m2 by the CKD-EPI equation at the screening visit. One repeat measurement is allowed.

* Inclusion Criteria for Healthy Adult Participants (Groups D):.
* Healthy adult participants must be 19 to 55 years of age, inclusive.

  i) Participants with any ethnicity can be included.

ii) Must have a BMI of 18.0 to 32.0 kg/m2 (inclusive), at the time of signing the ICF.

iii) Must have an eGFR of ≥ 90 mL/min/1.73m2 by the CKD-EPI equation at the screening visit. One repeat measurement is allowed.

Exclusion Criteria

- Exclusion Criteria for All Participants (Groups A, B, C, and D):.

i) Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.

ii) History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.

iii) Participant has a history of syncope and/or symptomatic orthostatic hypotension in the year prior to Day 1.

iv) History of cancer that has not been in full remission for >5 years (except basal cell skin cancer or squamous cell skin cancer with history of curative treatment and no recurrence for > 1 year prior to the screening visit).

* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 28 days post last dose
  Part 1
Number of participants with Serioues AEs (SAEs) | Up to 28 days post last dose
  Part 1
Number of participants with vital sign abnormalities | Up to 28 days post last dose
  Part 1
Body weight | Up to 28 days post last dose
  Part 1
Number of participants with 12-lead electrocardiogram abnormalities | Up to 28 days post last dose
  Part 1
Number of participants with physical examination abnormalities | Up to 28 days post last dose
  Part 1
Number of participants with clinical laboratory assessment abnormalities | Up to 28 days post last dose
  Part 1
Columbia-Suicide Severity Rating Scale (C-SSRS) | On Day 30
  Part 1
Maximum observed plasma concentration (Cmax) | Up to Day 29
  Part 2
Time of maximum observed plasma concentration (Tmax) | Up to Day 29
  Part 2
Area under the concentration-time curve in 1 dosing interval (AUC(TAU)) | Up to Day 29
  Part 2
Area under the plasma concentration-time curve from time zero to 24 hours (AUC(0-24)) | Up to Day 29
  Part 2
Apparent total body clearance (CLT/F) | Up to Day 29
  Part 2
Apparent volume of distribution (Vz/F) | Up to Day 29
  Part 2
Terminal elimination half-life (T-HALF) | Up to Day 29
  Part 2

SECONDARY OUTCOMES:
Cmax | Up to Day 29
  Part 1
Tmax | Up to Day 29
  Part 1
AUC(0-24) | Up to Day 29
  Part 1
AUC(TAU) | Up to Day 29
  Part 1
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to Day 29
  Part 1
CLT/F | Up to Day 29
  Part 1
Vz/F | Up to Day 29
  Part 1
T-HALF | Up to Day 29
  Part 1
Number of participants with AEs | Up to 28 days post last dose
  Part 2
Number of participants with SAEs | Up to 28 days post last dose
  Part 2
Number of participants with vital sign abnormalities | Up to 28 days post last dose
  Part 2
Body weight | Up to 28 days post last dose
  Part 2
Number of participants with 12-lead electrocardiogram abnormalities | Up to 28 days post last dose
  Part 2
Number of participants with physical examination abnormalities | Up to 28 days post last dose
  Part 2
Number of participants with clinical laboratory assessment abnormalities | Up to 28 days post last dose
  Part 2
C-SSRS | On Day 30
  Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Cenexel ACT (Anaheim Clinical Trials), Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com